CLINICAL TRIAL: NCT07252427
Title: Gut Microbial Characteristics in Patients With Comorbid Inflammatory Bowel Disease and Depressive Disorder
Brief Title: Gut Microbiota in IBD With Comorbid Depressive Disorder
Status: Recruiting | Type: Observational
Sponsor: Fang Tang (Other)
Responsible Party: Sponsor-Investigator, Fang Tang, Doctor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2024 (143)
Record Dates: First submitted 2025-11-16; First posted 2025-11-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-01

CONDITIONS: Inflammatory Bowel Disease; Depressive Disorder
Keywords: Inflammatory Bowel Disease; Depressive Disorder; Comorbidity; Gut Microbiome; Metabolomics
MeSH Terms: conditions — Inflammatory Bowel Diseases; Depressive Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples (2-5g), blood samples (2-5ml), and intestinal mucosal biopsy samples collected during routine medical examination and stored at -80°C for subsequent microbiome and metabolomics analyses.

GROUPS / COHORTS (3):
- IBD with Depressive Disorder Group
  Interventions: Other: Not applicable- observational study
- IBD without Depressive Disorder Group
  Interventions: Other: Not applicable- observational study
- Control Group
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — observational study with no assigned intervention

SUMMARY:
Inflammatory bowel disease (IBD) is often comorbid with depressive disorder, and the development and progression of both conditions are closely related to the composition of gut microbiota and metabolites. However, studies investigating their comorbidity using microbiome and metabolomics approaches remain limited.

This study aims to investigate the diversity changes in the gut microbiome and metabolome of patients with comorbid IBD and depressive disorder through multi-omics approaches, to identify specific microbial and metabolic signatures associated with the comorbidity of these two conditions, and to provide a molecular basis for elucidating the underlying mechanisms.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic inflammatory disorder of the gastrointestinal tract that significantly impairs patients' quality of life. Depressive disorder is a common comorbidity in patients with IBD, and the coexistence of the two conditions can exacerbate disease burden and complicate treatment management. Increasing evidence suggests that both IBD and depressive disorder are closely related to alterations in the gut microbiome and metabolome; however, studies focusing on the comorbidity of these two conditions using multi-omics approaches remain limited.

This cross-sectional observational study aims to investigate the diversity and compositional changes of the gut microbiome and metabolome in patients with comorbid IBD and depressive disorder. Fecal, blood, and intestinal mucosal samples will be collected from three groups: (1) patients with IBD and comorbid depressive disorder, (2) patients with IBD without depressive disorder, and (3) control group. Through multi-omics analysis, the study seeks to identify specific microbial taxa and metabolites associated with the comorbidity of IBD and depressive disorder, uncover differential microbial and metabolic profiles among the three groups, and explore the potential molecular mechanisms underlying the interaction between intestinal inflammation and depressive symptoms. The findings are expected to provide a scientific basis for the development of novel diagnostic biomarkers and therapeutic strategies for IBD patients with comorbid depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

IBD with Depressive Disorder Group:

1. Patients diagnosed with inflammatory bowel disease (ICD-10 codes: K50-K51).
2. History of depressive disorder diagnosis or previous use of antidepressant medications.
3. Age ≥ 18 years.
4. Willingness to participate and provision of written informed consent.

IBD without Depressive Disorder Group:

1. Patients diagnosed with inflammatory bowel disease (ICD-10 codes: K50-K51).
2. No history of depressive disorder diagnosis
3. No previous use of antidepressant medications.
4. Age ≥ 18 years.
5. Willingness to participate and provision of written informed consent.

Control Group:

1. No history of inflammatory bowel disease, depressive disorder, or use of antidepressant medications.
2. No gastrointestinal symptoms (e.g., diarrhea, constipation, abdominal pain) within the past 3 months, and no history of gastrointestinal diseases.
3. Age ≥ 18 years.
4. Willingness to participate and provision of written informed consent.

Exclusion Criteria:

1. Presence of other major chronic diseases or infections (e.g., malignancy, hypertension, diabetes, coronary heart disease).
2. Use of antibiotics or probiotic supplements within the past 6 months.
3. Inability or difficulty in providing biological samples.
4. Missing essential patient information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel disease with or without comorbid depressive disorder, and control participants, recruited from the First Affiliated Hospital of Shandong First Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-16 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota composition and relative abundance | Baseline
  The primary outcome is the expression level and diversity of gut microbial taxa identified through metagenomic analysis among the three study groups.

SECONDARY OUTCOMES:
Metabolite profiles and relative abundance | Baseline
  The secondary outcome is the expression level and diversity of serum and fecal metabolites identified through untargeted metabolomics analysis, and their correlations with gut microbial composition.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China